CLINICAL TRIAL: NCT05364463
Title: Randomized Clinical Trial on the Effect of Reactive Hyperemia and Ultrasound-guided Puncture on the Success Rate of Radial Artery Cannulation in Patients Undergoing Cardiac Catheterization
Brief Title: Effect of Reactive Hyperemia and Ultrasound-guided Puncture on the Success Rate of Radial Artery Cannulation (RadialHUS)
Acronym: RadialHUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EC093-21_FJD
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Myocardial Ischemia; Cardiac Catheterization
Keywords: Radial Artery; Hyperemia; Ultrasonography
MeSH Terms: conditions — Myocardial Ischemia; Hyperemia | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ultrasound and hyperemia (Experimental): Use of ultrasound and hyperemia to puncture radial artery.
  Interventions: Procedure: Methods for cannulating the radial artery in a cardiac catheterization
- Ultrasound only (Experimental): Use of ultrasound only to puncture radial artery.
  Interventions: Procedure: Methods for cannulating the radial artery in a cardiac catheterization
- Hyperemia only (Experimental): Use of hyperemia and palpation to puncture radial artery.
  Interventions: Procedure: Methods for cannulating the radial artery in a cardiac catheterization
- Palpation (No Intervention): Use of palpation to puncture radial artery (control group).

INTERVENTIONS:
Procedure: Methods for cannulating the radial artery in a cardiac catheterization — The puncture will be performed in each participant according to the method has been assigned randomly: ultrasound and hyperemia, ultrasound only, hyperemia only, palpation.
  Arms: Hyperemia only; Ultrasound and hyperemia; Ultrasound only

SUMMARY:
Aims: to evaluate the success rate of radial artery cannulation in patients undergoing cardiac catheterization, using different methods such as palpation, hyperemia or ultrasound-guided puncture, together or each method separately. Specifically, the success rate at the first attempt, the number of attempts with each technique and the time spent will be assessed.

The hypothesis is that there are different success rates for each puncture technique when cannulating radial artery for cardiac catheterization.

Methods: randomized clinical trial with four parallel groups, with operator blinding. Those patients who will have the radial artery cannulated for an interventional cardiology procedure will be selected.

Once the participant agrees to be included in the study and signs the informed consent, they are randomized to one of four groups: ultrasound and hyperemia puncture, only ultrasound puncture, only hyperemia puncture, palpation puncture (control group). Subsequently, an ultrasound assessment of the participant's radial artery (diameter, depth and systolic peak velocity) will be performed. Once in the intervention room, the puncture will be performed according to the corresponding method. The puncturing operator in charge will not perform the randomization or the ultrasound assessment to avoid bias.

Variables will be collected in an ad hoc questionnaire designed to respond all study aims. Regarding the sample size, accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 92 subjects per group are required to detect significant differences. Therefore, the total sample size would be made up of 368 participants, estimating losses of 5%.

For variables description and hypotheses contrast, the statistical program SPSS version 22.0 for Windows will be used, working with a significance level of 5%.

DETAILED DESCRIPTION:
Background: ultrasound-guided puncture seems to facilitate cannulation of the radial artery in patients who undergoing cardiac catheterization. The efficacy of reactive hyperemia has also been seen, however, the combination of different methods in radial artery puncture has not been evaluated.

Aims: to evaluate the success rate of radial artery cannulation in patients undergoing cardiac catheterization, using different methods such as palpation, hyperemia or ultrasound-guided puncture, together or each method separately. Specifically, success rate at the first attempt, attempts numbers with each technique and time spent will be assessed. Possible complications and perceived pain by the participant in each technique will be evaluated.

The hypothesis is that there are different success rates for each puncture technique when cannulating radial artery for cardiac catheterization.

Methods: randomized clinical trial with four parallel groups, with operator blinding.

Participation in the clinical trial does not imply an increased risk for the patient since both ultrasound and hyperemia are harmless and non-invasive methods.

Once the participant agrees to be included in the study and signs the informed consent, they are randomized to one of four groups: ultrasound and hyperemia puncture (for hyperemia, a blood pressure cuff is inflated 50mmHg above systolic until a maximum of 200mmHg for 5 minutes before puncture, it is known that maximum hyperemia is achieved 60 to 180 seconds after deflation), ultrasound puncture only, hyperemia puncture only, palpation puncture (control group).

Similarly, before the puncture, an ultrasound assessment of the participant's radial artery (diameter, depth and systolic peak velocity) will be performed. Once in the intervention room, the puncture will be performed according to the corresponding method. The puncturing operator will not perform the randomization or the ultrasound assessment to avoid bias.

Participation in the study ends once the radial artery has been cannulated with the guide according to the Seldinger technique.

The randomization sequence was generated by the center's Biostatistics and Epidemiology Unit. The four possible puncture methods were stratified by operator.

All operators have performed hundreds of radial punctures by palpation and more than 20 ultrasound-guided punctures, as established by the study of the learning curve carried out by Jayanti S et al, before starting participants recruitment.

All the variables will be collected in an ad hoc questionnaire designed to respond all study objectives.

Regarding the sample size, accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 92 subjects per group are required to detect a statistically significant difference, which for the control group (traditional puncture) is expected to be 0.44 the percentage of success at the first puncture attempt, and for the rest is at least 0.65. Therefore, the total sample size would be made up of 368 participants, estimating a follow-up loss of 5%.

Regarding the statistical analysis, the quantitative variables will be described with the mean and the standard deviation if they follow a normal distribution, or with the median and the interquartile range if they do not follow a normal distribution. The normality will be contrasted using the Kolmogorov-Smirnov test. The qualitative variables will be described through the distribution of frequencies and percentages.

For the comparisons of the quantitative variables following a normal distribution, the one factor analysis of variance (ANOVA) will be used for the global comparison, and the Student's t-test in the comparisons by pairs. For variables do not following a normal distribution, the Kruskal Wallis test will be used in the global comparison, and Dunn's test in pairwise comparisons. For comparisons of qualitative variables, the Chi-square test will be used, or Fisher's exact test in those situations in which the criteria for using the Chi-square are not met. In pairwise comparisons, the Bonferroni correction will be applied for multiple comparisons.

In all hypothesis contrasts, a significance level of 5% will be used. The statistical program SPSS version 22.0 for Windows will be used.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* understand, accept and sign the informed consent
* participants undergoing radial artery cannulation for a diagnostic, therapeutic, or structural interventional cardiology procedure
* patent radial artery in the previous ultrasound evaluation

Exclusion Criteria:

* systolic blood pressure greater than 150mmHg
* diagnosis of acute myocardial infarction (with or without ST-segment elevation)
* previous surgeries that have affected the arterial system of the upper limbs (arteriovenous fistula, radial artery for bypass surgery, etc.)
* language barrier that hinders a clear study understanding for potential participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of success at first puncture attempt | During radial artery puncture, it will be assessed whether cannulation can be achieved at the first attempt
  It is assessed whether the radial artery is cannulated in the first puncture without removing the needle from the skin
Number of punctures | During radial artery cannulation, punctures number have been necessary will be measured
  The punctures number have been necessary to achieve radial artery cannulation will be measured
Time to cannulate | During radial artery cannulation, the time will be measured from the needle is inserted into the skin for the first time until the guidewire enters the arterial lumen, stopping time when the needle is out of the skin (if more than one puncture)
  The time in minutes and seconds has been necessary to cannulate radial artery will be measured

SECONDARY OUTCOMES:
Rate of possible complications | During or just after the cardiac catheterization, the possible complications related to the arterial puncture will be assessed
  Complications that may arise after arterial puncture such as spasm, hematoma, cyanosis, coldness, paresthesia, etc.
Perceived pain | The perceived pain will be recorded at the end of the radial artery cannulation
  The perceived pain by the patient will be recorded on a 0 to 10 scale, with 0 being no pain and 10 being the maximum possible imagined pain

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Sánchez, RN, BsC, MSc, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (1):
- Fundación Jiménez Díaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
After completing the recruitment, the data collected will be analyzed for publication

REFERENCES:
- [Background] Deftereos S, Giannopoulos G, Kossyvakis C, Driva M, Kaoukis A, Raisakis K, Theodorakis A, Panagopoulou V, Lappos S, Tampaki E, Pyrgakis V, Stefanadis C. Radial artery flow-mediated dilation predicts arterial spasm during transradial coronary interventions. Catheter Cardiovasc Interv. 2011 Apr 1;77(5):649-54. doi: 10.1002/ccd.22688. PMID 20549693
- [Background] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671
- [Background] Doubell J, Kyriakakis C, Weich H, Herbst P, Pecoraro A, Moses J, Griffiths B, Snyman HW, Kabwe L, Du Toit R, Joubert L, Hassan K, Doubell A. Radial artery dilatation to improve access and lower complications during coronary angiography: the RADIAL trial. EuroIntervention. 2021 Mar 19;16(16):1349-1355. doi: 10.4244/EIJ-D-19-00207. PMID 31746742
- [Background] Thijssen DHJ, Bruno RM, van Mil ACCM, Holder SM, Faita F, Greyling A, Zock PL, Taddei S, Deanfield JE, Luscher T, Green DJ, Ghiadoni L. Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans. Eur Heart J. 2019 Aug 7;40(30):2534-2547. doi: 10.1093/eurheartj/ehz350. PMID 31211361
- [Background] Lanza GA, Cesarano M, De Vita A, Villano A, Milo M, Russo G, Crea F. Effect of Remote Ischemic Preconditioning on Coronary Procedure-Related Impairment of Vascular Dilator Function. J Am Coll Cardiol. 2016 Dec 6;68(22):2490-2492. doi: 10.1016/j.jacc.2016.08.071. No abstract available. PMID 27908357
- [Background] Seto AH, Roberts JS, Abu-Fadel MS, Czak SJ, Latif F, Jain SP, Raza JA, Mangla A, Panagopoulos G, Patel PM, Kern MJ, Lasic Z. Real-time ultrasound guidance facilitates transradial access: RAUST (Radial Artery access with Ultrasound Trial). JACC Cardiovasc Interv. 2015 Feb;8(2):283-291. doi: 10.1016/j.jcin.2014.05.036. Epub 2015 Jan 14. PMID 25596790
- [Background] Jayanti S, Juergens C, Makris A, Hennessy A, Nguyen P. The Learning Curves for Transradial and Ultrasound-Guided Arterial Access: An Analysis of the SURF Trial. Heart Lung Circ. 2021 Sep;30(9):1329-1336. doi: 10.1016/j.hlc.2021.02.006. Epub 2021 Mar 12. PMID 33722490
- See also: ESC Guidelines — http://www.revespcardiol.org/es-pdf-S0300893218306377